CLINICAL TRIAL: NCT06128759
Title: The Effect of Focusing on the Maryam's Flower During the Birth Process on Labor Pain, Labor Duration and Perceived Fatigue in Birth
Brief Title: Focusing on the Maryam's Flower During the Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sümeyye BAL, Ph.D., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/294
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maryam's Flower Group (Experimental): Maryam's flower will place in a bowl of water and left in the room of the pregnant women who will at 1 cm cervical dilatation and in the first phase of the labor. It will explain to the pregnant women that the leaves of the plant would open up in the water, and they will ask to imagine that the birth canal would simultaneously open up. In effect, they will told to focus on the opening of these leaves during the course of the labor.. After birth, the flower used only as a focusing method will be removed from the water and its water will be poured.
  Interventions: Other: Focusing on Maryam's Flower
- control group (No Intervention): will provided with standard midwifery care.

INTERVENTIONS:
Other: Focusing on Maryam's Flower — Effect of Focusing on Maryam's Flower During the First Phase of the labor
  Other Names: Foccusing on Maryam's Flower
  Arms: Maryam's Flower Group

SUMMARY:
To determine the Effect of Focusing on the Virgin Mary Flower during the Birth Process on Labor Pain, Labor Duration and Perceived Fatigue in Birth.

Method: The study will be completed in a randomized controlled manner with a total of 126 primiparous pregnant women, 63 in the experimental group and 63 in the control group. Pregnant women in the experimental group will focus on the Virgin Mary flower in the water-filled jar and imagine that their uterus and birth path are opening like the branches of the Virgin Mary flower that blooms as labor pains come. There will be no intervention in the control group other than routine midwifery care. Research data will be collected with the Pregnant Introduction and Birth Process Follow-up Form, Visual Analog Scale, and Visual Similarity Scale for Fatigue.

DETAILED DESCRIPTION:
Design and Settings: This randomized controlled experimental study will conducted in the delivery room of the, Turkey between the dates of November 2023 and April 2024

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* being in 37-42 weeks of pregnancy,
* being primiparous,
* having a single healthy fetus,
* cervical dilatation not more than 3 cm.the one which,
* in the first stage of labor,
* Does not have any complications preventing vaginal birth,
* volunteer women who do not have disabilities in communication and perception

Exclusion Criteria:

* maternal and fetal complications
* pregnant with assisted reproductive techniques,
* having a presentation anomaly,
* having a twin pregnancy,
* electing cesarean section,
* Women whose cervical dilatation exceeds 3 cm and who are not willing to participate in the study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
severity of labor pain by VAS | immediately after intervention
  Visual Analog Scale: The scale features a 10-cm long vertical line, with 0 at the bottom end and 10 at the top end
Visual Similarity Scale for Fatigue | immediately after intervention
  The scale consists of two subscales, fatigue and energy, and 18 items. There are 10 cm long horizontal lines with positive expressions at one end and negative expressions at the other end of the YİBGS. While the items of the fatigue subscale progress from positive to negative, the energy subscale has the opposite order. The lowest score obtained from the fatigue subscale is 0 and the highest score is 130. In the energy subscale, scores range from 0 to 50.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye BAL, Study Chair — Ondokuz Mayıs University; Sümeyye BAL, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No